CLINICAL TRIAL: NCT00886210
Title: Clinical Impact of Routine Abdominal Drainage After Laparoscopic Cholecystectomy. A Prospective Randomized Study
Brief Title: Clinical Impact of Routine Abdominal Drainage After Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Mansoura University, Mansoura University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: abdominal drainage
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Abdominal Drainage; Laparoscopic Cholecystectomy; Gall Stones
Keywords: drain; laparoscopic cholecystectomy; pneumoperitonum
MeSH Terms: conditions — Gallstones | interventions — Drainage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1LC with drain (Active Comparator): Under general anesthesia, and same antibiotics (3rd generation cephalosporin). Surgery was performed using conventional four ports umbilical port, port below xiphoid and two ports below right costal margin. Pneumoperitonum at pressure 12 mmHg. In group A nelton catheter (no 20) inserted at the end of operation.
  Interventions: Procedure: intra abdominal drain
- 2LC without drain (Active Comparator): Under general anesthesia, and same antibiotics (3rd generation cephalosporin). Surgery was performed using conventional four ports umbilical port, port below xiphoid and two ports below right costal margin. Pneumoperitonum at pressure 12 mmHg. no drain at the end of operation.
  Interventions: Procedure: LC without drain

INTERVENTIONS:
Procedure: intra abdominal drain — Under general anesthesia, and same antibiotics (3rd generation cephalosporin). Surgery was performed using conventional four ports umbilical port, port below xiphoid and two ports below right costal margin. Pneumoperitonum at pressure 12 mmHg. In group A nelton catheter (no 20) inserted at the end of operation.
  Other Names: Group A
  Arms: 1LC with drain
Procedure: LC without drain — Under general anesthesia, and same antibiotics (3rd generation cephalosporin). Surgery was performed using conventional four ports umbilical port, port below xiphoid and two ports below right costal margin. Pneumoperitonum at pressure 12 mmHg. In group no drain at the end of operation.
  Other Names: Group B
  Arms: 2LC without drain

SUMMARY:
Patients and methods: 100 patients were included in this study. They divided into two groups, group (A) with drain and group (B) without drain. The investigators recorded the effect of drainage on, postoperative pain (Po-P) using visual analogue scale VAS at 6, 24, 48 hours and 1 week postoperative nausea/vomiting at 6, 24, 48 hours postoperative, abdominal collection, hospital stay, chest complication, and postoperative body temperature.

DETAILED DESCRIPTION:
The patients were randomized into two groups using enclosed envelope. Group (A) with drain included 50 patients, and group (B) without drain included 50 patients.

Under general anesthesia, and same antibiotics (3rd generation cephalosporin) Surgery was performed using conventional four ports umbilical port, port below xiphoid and two ports below right costal margin. Pneumoperitonum at pressure 12 mmHg. In group A nelton catheter (no 20) was inserted at the end of operation.

The Intraoperative parameter observed included duration of the operation, amount of CO2 used in the operation, bile escape, saline irrigation during operation and volume of blood loss were recorded.

The patients started oral feeding 8 hours (h) postoperatively; abdominal ultrasound was done for all patients in both groups on day of discharge to show any collection or free fluid in the abdomen. The patients were usually discharged after removal of drain, and when the patient surgically free.

Postoperative pain was evaluated at 6 h, 24 h, 48, 1 week after operation using a visual analog scale (VAS) with which each patients noted the severity of pain at each evaluated time using a linear between zero (no pain) and 10 (severe pain). Postoperative analgesia in the form of non steroidal anti-inflammatory drug (NSAID) was administered intramuscularly when required. If the patients still complained of pain and required strong analgesic, (1 mg/kg pethidine intramuscularly) was administered. The total dose of these medications were recorded.

Postoperative maximum body temperatures were recorded at (6 h, 24 h, and 48 h) for all patients.

PONV were assessed postoperative after 6 h, 24 h and after 48 h. Metocloprpamide was given if the patients required reduction of nausea and the total dose of this medication was recorded. The frequency of vomiting was recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients with gallbladder stones and laparoscopic cholecystectomy

Exclusion Criteria:

* patients above 80 years old
* patients with acute cholecystitis
* patients with history of upper laparotomy
* patients with a hemorrhagic tendency due to cirrhosis
* patients refused to give informed consent and patients who were converted to open cholecystectomy

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
pain, nausea and vomiting | 30 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Elnakeeb, MD, Principal Investigator — Mansoura University Hospital
Locations (1):
- Ayman Elnakeeb, Al Mansurah, Egypt

REFERENCES:
- [Result] Hawasli A, Brown E. The effect of drains in laparoscopic cholecystectomy. J Laparoendosc Surg. 1994 Dec;4(6):393-8. doi: 10.1089/lps.1994.4.393. PMID 7881142
- [Result] Uchiyama K, Tani M, Kawai M, Terasawa H, Hama T, Yamaue H. Clinical significance of drainage tube insertion in laparoscopic cholecystectomy: a prospective randomized controlled trial. J Hepatobiliary Pancreat Surg. 2007;14(6):551-6. doi: 10.1007/s00534-007-1221-x. Epub 2007 Nov 30. PMID 18040619
- See also: Mansoura university hospital — http://home.mans.eun.eg/